CLINICAL TRIAL: NCT05563714
Title: Anticoagulation With Enhanced Gastrointestinal Safety (AEGIS): A Pragmatic Randomized Trial to Evaluate Clinician Outreach to Reduce Upper Gastrointestinal Bleeding Risk in Patients Taking Warfarin and Antiplatelet Therapy
Brief Title: Anticoagulation With Enhanced Gastrointestinal Safety
Acronym: AEGIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jacob E Kurlander, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00217771; K23DK118179 (NIH)
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Upper Gastrointestinal Bleeding; Peptic Ulcer Hemorrhage; Anticoagulant-induced Bleeding
Keywords: Warfarin; Proton pump inhibitor; Antiplatelet therapy; Gastroprotection; Aspirin; Thienopyridine; Patient safety; Anticoagulation
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Peptic Ulcer Hemorrhage

STUDY DESIGN:
Intervention Model Description: Randomization (1:1) of clinicians and patients to CNNF vs. wait list control will be done at the cluster level according to the identity of the clinician to be contacted. Clinician randomization will be stratified by number of eligible patients, and by procedural vs. non-procedural specialty. Randomization will be carried out by the study statistician. For each included clinician, up to 4 patients will be included in their cluster. If a clinician is selected to participate who has more than 4 eligible patients, 4 of their patients will be randomly selected to participate.
Masking Description: Neither patients, clinicians, or anticoagulation staff can practically be blinded. We will attempt to blind the research staff who are making patient calls at week 7-10 to the randomization group of the patient by not providing them with any information that would allow them to infer the randomization group, by not having them enter the electronic health record for the patients, where such information could be obtained, and by excluding any information from the call script that might help identify the randomization group. However, if due to staffing or personnel issues, blinded research staff are unable to complete all patient calls within the specified time frame, unblinded research staff will assist with completing patient calls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinician Notification with Nurse Facilitation (CNNF) (Experimental)
  Interventions: Behavioral: Clinician Notification with Nurse Facilitation (CNNF)
- Wait List Control (Usual care) (Other)
  Interventions: Behavioral: Wait list control

INTERVENTIONS:
Behavioral: Clinician Notification with Nurse Facilitation (CNNF) — An anticoagulation clinic nurse sends a templated message to the patient's target clinician that identifies the patient as high risk for upper GI bleeding, summarizes guidelines on appropriate antiplatelet medication use and PPI gastroprotection, and recommends that the clinician consider either discontinuing the patient's antiplatelet medication(s) or initiating a PPI for gastroprotection. The nurse will also offer to pend the order for a PPI if the clinician wants to initiate a PPI and will provide education to the patient on any medication changes recommended by the clinician.
  Arms: Clinician Notification with Nurse Facilitation (CNNF)
Behavioral: Wait list control — The anticoagulation clinic will not send the clinician notification letter or other project-specific materials to the clinician or patient, and the patient will be included on a list of patients who will receive the intervention at the conclusion of the trial.
  Arms: Wait List Control (Usual care)

SUMMARY:
This study is a pragmatic cluster randomized controlled trial to evaluate the effectiveness of a clinician-facing implementation strategy on the use of medication optimization (defined as either discontinuation of all antiplatelet therapy or initiation of and adherence to a proton pump inhibitor (PPI)) to reduce upper GI bleeding risk in patients prescribed anticoagulant-antiplatelet therapy (AAT) relative to usual care.

DETAILED DESCRIPTION:
This is a pragmatic, single-center cluster randomized controlled trial to evaluate a clinician-facing implementation strategy to increase the use of evidence-based practices (EBPs) to reduce bleeding in patients who are using AAT and who are managed by the Michigan Medicine anticoagulation monitoring service. The active intervention is clinician notification with nurse facilitation (CNNF), which consists of an anticoagulation clinic nurse sending an electronic health record message that identifies the patient as high risk for upper GI bleeding and recommends either discontinuing the antiplatelet agent or initiating a PPI; the nurse also pends medication orders for PPIs and provides patient education upon request. Clinicians will be cluster randomized, such that up to 4 patients cared for by each clinician will receive the same clinician-level notification.

This study will use a "wait-listed design," in which patients will be randomized to either have their clinicians receive CNNF or be included in a wait-list control group. At the completion of the study, the patients who were randomized to the wait-list control group will receive the intervention.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Enrollment with the Michigan Medicine anticoagulation monitoring service
* Currently prescribed warfarin with anticipated use for ≥90 days on day 1 of trial enrollment, according to the electronic health record documentation.
* Currently prescribed an antiplatelet medication (aspirin, clopidogrel, ticagrelor, or prasugrel) according to the electronic health record medication list

Inclusion Criteria for Clinicians:

* Cardiologists at Michigan Medicine who in the prior year had a face-to-face or virtual visit with a patient who meets eligibility criteria
* Michigan Medicine primary care providers for patients who meet eligibility criteria
* Clinicians in any specialty who are designated as the clinician of record with the anticoagulation clinic for a patient who meets eligibility criteria

Exclusion Criteria for Patients:

* Age less than 18
* Currently prescribed a PPI
* Documented intolerance or allergy to PPI use
* Left ventricular assist device
* Heart transplant
* Participation in a previous pilot study of these implementation strategies

Exclusion Criteria for Clinicians:

* Cardiologists specializing in electrophysiology or who saw the patient for a clinic visit related to a TAVI procedure unless they are the clinician of record for a patient followed by the anticoagulation service who does not have a Michigan Medicine PCP.
* Participation in a previous pilot study of these QI strategies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob E Kurlander, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Arm - Clinician Notification With Nurse Facilitation (CNNF); Clinician Arm - Clinician Notification With Nurse Facilitation (CNNF): Clinician Notification with Nurse Facilitation (CNNF): An anticoagulation clinic nurse sends a templated message to the patient's target clinician that identifies the patient as high risk for upper GI bleeding, summarizes guidelines on appropriate antiplatelet medication use and PPI gastroprotection, and recommends that the clinician consider either discontinuing the patient's antiplatelet medication(s) or initiating a PPI for gastroprotection. The nurse will also offer to pend the order for a PPI if the clinician wants to initiate a PPI and will provide education to the patient on any medication changes recommended by the clinician.
- Patient Arm - Wait List Control (Usual Care); Clinician Arm - Wait List Control (Usual Care): Wait list control: The anticoagulation clinic will not send the clinician notification letter or other project-specific materials to the clinician or patient, and the patient will be included on a list of patients who will receive the intervention at the conclusion of the trial.
Period: Overall Study
Arm/Group | Patient Arm - Clinician Notification With Nurse Facilitation (CNNF) | Patient Arm - Wait List Control (Usual Care) | Clinician Arm - Clinician Notification With Nurse Facilitation (CNNF) | Clinician Arm - Wait List Control (Usual Care)
Started | 110 | 110 | 61 | 60
Completed | 81 | 83 | 61 | 60
Not Completed | 29 | 27 | 0 | 0
Not completed — Death | 2 | 2 | 0 | 0
Not completed — Patient unenrollment from Anticoagulation Monitoring Service prior to primary outcome assessment | 4 | 3 | 0 | 0
Not completed — Patient medication change - warfarin discontinuation, switch to DOAC therapy | 1 | 2 | 0 | 0
Not completed — Patient hospitalized for entirety of primary outcome assessment timeframe | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 22 | 19 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Arm - Clinician Notification With Nurse Facilitation (CNNF) | Patient Arm - Wait List Control (Usual Care) | Clinician Arm - Clinician Notification With Nurse Facilitation (CNNF) | Clinician Arm - Wait List Control (Usual Care) | Total
Number analyzed (Participants) | 110 | 110 | 61 | 60 | 341
Age, Customized [Mean (Standard Deviation); unit: years] — Population: This data was not collected for clinician participants.
  years
    Patient Characteristics - Age: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Patient Characteristics - Age | 61 (16) | 62 (15) |  |  | 62 (15)
Age, Customized [Median (Inter-Quartile Range); unit: years] — Population: This data was not collected for clinician participants.
  years
    Patient Characteristics - Age: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Patient Characteristics - Age | 64 [52 to 73] | 65 [52 to 74] |  |  | 64 [52 to 73]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Patient and clinician data are reported separately.
  Participants
    Patient Characteristics - Sex: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Patient Characteristics - Sex: Female | 43 | 36 |  |  | 79
    Patient Characteristics - Sex: Male | 67 | 74 |  |  | 141
    Clinician Characteristics - Sex: number analyzed (Participants) | 0 | 0 | 61 | 60 | 121
    Clinician Characteristics - Sex: Female |  |  | 26 | 23 | 49
    Clinician Characteristics - Sex: Male |  |  | 35 | 37 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This data was not collected for clinician participants.
  Participants
    number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Hispanic or Latino | 1 | 1 |  |  | 2
    Not Hispanic or Latino | 108 | 104 |  |  | 212
    Unknown or Not Reported | 1 | 5 |  |  | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This data was not collected for clinician participants.
  Participants
    number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    American Indian or Alaska Native | 1 | 0 |  |  | 1
    Asian | 4 | 1 |  |  | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Black or African American | 15 | 6 |  |  | 21
    White | 86 | 99 |  |  | 185
    More than one race | 0 | 0 |  |  | 0
    Unknown or Not Reported | 4 | 4 |  |  | 8
Region of Enrollment [Number; unit: participants]
  United States | 110 | 110 | 61 | 60 | 341
Antiplatelet Therapy [Count of Participants; unit: Participants] — Population: This data was not collected for clinician participants.
  Participants
    number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Aspirin | 105 | 96 |  |  | 201
    Clopidogrel | 4 | 12 |  |  | 16
    Dual Antiplatelet Therapy | 1 | 2 |  |  | 3
Concomitant Medications [Count of Participants; unit: Participants] — Population: This data was not collected for clinician participants.
  Participants
    H2 Receptor Antagonist Use: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    H2 Receptor Antagonist Use | 11 | 5 |  |  | 16
    Oral Non-Steroidal Anti-Inflammatory Drug (NSAID) Use: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Oral Non-Steroidal Anti-Inflammatory Drug (NSAID) Use | 2 | 2 |  |  | 4
    Selective Serotonin Reuptake Inhibitor (SSRI) Use: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Selective Serotonin Reuptake Inhibitor (SSRI) Use | 17 | 11 |  |  | 28
    Oral Glucocorticoid Use: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Oral Glucocorticoid Use | 5 | 5 |  |  | 10
    Aldosterone Antagonist Use: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Aldosterone Antagonist Use | 22 | 17 |  |  | 39
Medical History [Count of Participants; unit: Participants] — Population: This data was not collected for clinician participants.
  Participants
    Atrial Fibrillation: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Atrial Fibrillation | 46 | 40 |  |  | 86
    Venous Thromboembolism: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Venous Thromboembolism | 34 | 28 |  |  | 62
    Valve Replacement: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Valve Replacement | 46 | 52 |  |  | 98
    Coronary Artery Disease: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Coronary Artery Disease | 43 | 48 |  |  | 91
    Antiphospholipid Syndrome: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Antiphospholipid Syndrome | 11 | 4 |  |  | 15
    Peripheral Artery Disease: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Peripheral Artery Disease | 20 | 17 |  |  | 37
    Cerebrovascular Disease: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Cerebrovascular Disease | 27 | 19 |  |  | 46
    GI Bleeding or Peptic Ulcer Disease: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    GI Bleeding or Peptic Ulcer Disease | 6 | 2 |  |  | 8
Clinician Specialty [Count of Participants; unit: Participants] — Population: As up to 4 patients were assigned to each clinician cluster, this data is reported separately for patient and clinician participants.
  Participants
    Patient Characteristics - Clinician Specialty: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Patient Characteristics - Clinician Specialty: Cardiology | 54 | 56 |  |  | 110
    Patient Characteristics - Clinician Specialty: Electrophysiology | 2 | 2 |  |  | 4
    Patient Characteristics - Clinician Specialty: Hematology | 3 | 3 |  |  | 6
    Patient Characteristics - Clinician Specialty: Hepatology | 0 | 1 |  |  | 1
    Patient Characteristics - Clinician Specialty: Primary Care | 33 | 28 |  |  | 61
    Patient Characteristics - Clinician Specialty: Pulmonology | 0 | 1 |  |  | 1
    Patient Characteristics - Clinician Specialty: Radiology | 4 | 1 |  |  | 5
    Patient Characteristics - Clinician Specialty: Rheumatology | 4 | 0 |  |  | 4
    Patient Characteristics - Clinician Specialty: Thoracic Surgery | 8 | 8 |  |  | 16
    Patient Characteristics - Clinician Specialty: Vascular Surgery | 2 | 10 |  |  | 12
    Clinician Characteristics - Clinician Specialty: number analyzed (Participants) | 0 | 0 | 61 | 60 | 121
    Clinician Characteristics - Clinician Specialty: Cardiology |  |  | 23 | 22 | 45
    Clinician Characteristics - Clinician Specialty: Electrophysiology |  |  | 1 | 1 | 2
    Clinician Characteristics - Clinician Specialty: Hematology |  |  | 2 | 2 | 4
    Clinician Characteristics - Clinician Specialty: Hepatology |  |  | 0 | 1 | 1
    Clinician Characteristics - Clinician Specialty: Primary Care |  |  | 27 | 25 | 52
    Clinician Characteristics - Clinician Specialty: Pulmonology |  |  | 0 | 1 | 1
    Clinician Characteristics - Clinician Specialty: Radiology |  |  | 2 | 1 | 3
    Clinician Characteristics - Clinician Specialty: Rheumatology |  |  | 1 | 0 | 1
    Clinician Characteristics - Clinician Specialty: Thoracic Surgery |  |  | 4 | 4 | 8
    Clinician Characteristics - Clinician Specialty: Vascular Surgery |  |  | 1 | 3 | 4
Clinician Proceduralist Status [Count of Participants; unit: Participants] — Population: As up to 4 patients were assigned to each clinician cluster, this data is reported separately for patient and clinician participants.
  Participants
    Patient Characteristics - Clinician Proceduralist Status: number analyzed (Participants) | 110 | 110 | 0 | 0 | 220
    Patient Characteristics - Clinician Proceduralist Status: Proceduralist | 16 | 21 |  |  | 37
    Patient Characteristics - Clinician Proceduralist Status: Non-Proceduralist | 94 | 89 |  |  | 183
    Clinician Characteristics - Clinician Proceduralist Status: number analyzed (Participants) | 0 | 0 | 61 | 60 | 121
    Clinician Characteristics - Clinician Proceduralist Status: Proceduralist |  |  | 8 | 9 | 17
    Clinician Characteristics - Clinician Proceduralist Status: Non-Proceduralist |  |  | 53 | 51 | 104
Years Since Medical School Completed [Mean (Standard Deviation); unit: years] — This measure applies only to Clinician participants. Population: This measure applies only to clinician participants and data was not collected for patient participants.
  years
    number analyzed (Participants) | 0 | 0 | 61 | 60 | 121
    (all) |  |  | 23 (12) | 23 (11) | 23 (11)
Years Since Medical School Completed [Median (Inter-Quartile Range); unit: years] — Population: This measure applies only to clinician participants and data was not collected for patient participants.
  years
    number analyzed (Participants) | 0 | 0 | 61 | 60 | 121
    (all) |  |  | 22 [14 to 30] | 22 [14 to 30] | 22 [14 to 30]

OUTCOME MEASURES:

1. Primary Outcome: ITT Analysis - Percent of Patients Reporting Medication Optimization
Description: The percent of patients reporting medication optimization is defined as the number of patients who either discontinue all antiplatelet medications (none in the past 7 days) or initiate and adhere to a proton pump inhibitor (PPI) (use for at least 5 of the prior 7 days) based on self-report at week 7-10 divided by the total number of patients in that randomization arm.
Time Frame: Up to 10 weeks
Population: All patients who entered the study were included in this intention-to-treat analysis. Multiple imputation was used to account for missing data for patients lost to follow-up, including patients who were closed to the anticoagulation service, discontinued warfarin therapy, died or were hospitalized throughout the data collection window, were unreachable by phone, declined to participate in the phone survey, or self-reported non-use of antiplatelet therapy or use of PPIs at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Arm - Clinician Notification With Nurse Facilitation (CNNF) | Patient Arm - Wait List Control (Usual Care)
Number analyzed (Participants) | 110 | 110
Participants
  Reached by phone & achieved medication optimization | 30 | 2
  Reached by phone & did not achieve medication optimization | 29 | 65
  Data Imputed - Reached by phone but reported non-use of antiplatelet therapy at baseline | 15 | 10
  Data Imputed - Reached by phone but reported use of or uncertain use of PPIs at baseline | 8 | 6
  Data Imputed - Patients lost to follow-up due to death or hospitalization | 2 | 3
  Data Imputed - Patients closed to the anticoagulation service or who discontinued warfarin therapy | 5 | 5
  Data Imputed - Patients unable to be reached by phone or who declined to participate in the survey | 21 | 19
Statistical Analysis 1: Comparison: Patient Arm - Clinician Notification With Nurse Facilitation (CNNF) vs Patient Arm - Wait List Control (Usual Care); Adjusted OR (base model), 95% CI - Includes clinician proceduralist vs non-proceduralist status as a co-variate; Test type: Superiority; p < 0.001, generalized linear mixed effects model; Odds Ratio (OR) = 5.22, 95% CI 2-sided [2.41 to 11.33] — Adjusted OR (base model)
Statistical Analysis 2: Comparison: Patient Arm - Clinician Notification With Nurse Facilitation (CNNF) vs Patient Arm - Wait List Control (Usual Care); Adjusted OR (expanded model), 95% CI - Adjusted for clinician proceduralist vs non-proceduralist status, patient age, sex, race, ethnicity, number of comorbidities, antiplatelet therapy used at baseline, and baseline use of H2 receptor antagonists; Test type: Superiority; p < 0.001, generalized linear mixed effects model; Odds Ratio (OR) = 5.76, 95% CI 2-sided [2.54 to 13.05] — Adjusted OR (expanded model)

2. Primary Outcome: Modified Completer Analysis - Percent of Patients Reporting Medication Optimization
Description: as for outcome 1
Time Frame: Up to 10 weeks
Population: Patients who self-reported either not using antiplatelet therapy or using a PPI at the start of the trial during the week 7-10 phone survey, and those who were lost to follow up were excluded from the modified completer analysis (n=94).
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Arm - Clinician Notification With Nurse Facilitation (CNNF) | Patient Arm - Wait List Control (Usual Care)
Number analyzed (Participants) | 59 | 67
Participants
  All patients who reported non-use of antiplatelet therapy or use of PPI gastroprotection | 30 | 2
  Stopped antiplatelet therapy | 17 | 1
  Started a PPI | 11 | 1
  Stopped antiplatelet therapy and started a PPI | 2 | 0
Statistical Analysis 1: Comparison: Patient Arm - Clinician Notification With Nurse Facilitation (CNNF) vs Patient Arm - Wait List Control (Usual Care); Adjusted OR (base model), 95% CI - Included clinician proceduralist vs non-proceduralist status as a co-variate; Test type: Superiority; p < 0.001, generalized linear mixed effects model; Odds Ratio (OR) = 29.3, 95% CI 2-sided [6.07 to 141.49] — Adjusted OR (base model)
Statistical Analysis 2: Comparison: Patient Arm - Clinician Notification With Nurse Facilitation (CNNF) vs Patient Arm - Wait List Control (Usual Care); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, generalized linear mixed effects model; Odds Ratio (OR) = 43.6, 95% CI 2-sided [6.56 to 289.88] — Adjusted OR (expanded model)

3. Secondary Outcome: ITT Analysis - Percent of Patients With Documented Recommendation Regarding Antiplatelet Therapy Cessation or PPI Initiation
Description: The number of patients who have a recommendation from a Michigan Medicine clinician to either discontinue all antiplatelet medications or initiate a PPI divided by the total number of patients in that randomization arm.
Time Frame: Up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Arm - Clinician Notification With Nurse Facilitation (CNNF) | Patient Arm - Wait List Control (Usual Care)
Number analyzed (Participants) | 110 | 110
Participants
  Received a recommendation for medication optimization | 75 | 1
  Received a recommendation to discontinue antiplatelet therapy | 32 | 1
  Received a recommendation to initiate a PPI | 38 | 0
  Received a recommendation to discontinue antiplatelet therapy and to initiate a PPI | 5 | 0
Statistical Analysis 1: Comparison: Patient Arm - Clinician Notification With Nurse Facilitation (CNNF) vs Patient Arm - Wait List Control (Usual Care); We used generalized linear mixed effects modeling (logit link) to estimate the odds of medication optimization at week 7-10. This model included fixed effects for CNNF (vs. usual care), target provider specialty and size, and a random effect for clinician to account for the clustering of patients. We report the log odds ratios with corresponding confidence intervals for the main effect. The main effect was tested at a two-sided 5% significance level; Test type: Superiority — Adjusted OR, 95% CI (base model) - Included clinician proceduralist vs non-proceduralist status as a co-variate; p < 0.001, generalized linear mixed effects model; Odds Ratio, log = 19.86, 95% CI 2-sided [10.63 to 29.09]

ADVERSE EVENTS:
Time Frame: Up to 10 weeks
Description: This study did not proactively monitor for adverse events as the trial constituted a quality improvement effort intended to improve the use of evidence-based practices, and decisions regarding changes in drug treatment were made as part of usual care. However, if any adverse events affecting patient participants were identified during data collection, they were documented in a database for regulatory review. No adverse events were assessed/monitored for clinician participant arms.
Arm/Group | Patient Arm - Clinician Notification With Nurse Facilitation (CNNF) | Patient Arm - Wait List Control (Usual Care) | Clinician Arm - Clinician Notification With Nurse Facilitation (CNNF) | Clinician Arm - Wait List Control (Usual Care)
All-Cause Mortality (participants affected / at risk) | 2/110 | 2/110 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/110 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/110 | 0/110 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT05563714/Prot_SAP_000.pdf